CLINICAL TRIAL: NCT05197062
Title: A Phase 1, Open Label Study to Characterize the Absorption, Metabolism, and Excretion of 14C JNJ-67953964 After a Single Dose in Healthy Adult Male Participants
Brief Title: A Study of 14C JNJ-67953964 in Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR109135; 2021-005130-42 (EudraCT Number); 67953964MDD1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-01-17; First posted 2022-01-19 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Aticaprant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 14C-aticaprant (Experimental): Participants in Group A (without duodenal fluid collection) and Group B (with duodenal fluid collection) will receive a single oral dose of 14C-aticaprant on Day 1.
  Interventions: Drug: 14C-aticaprant

INTERVENTIONS:
Drug: 14C-aticaprant — 14C-aticaprant will be administered orally as capsule on Day 1.
  Other Names: JNJ-67953964

SUMMARY:
The purpose of this study is to assess the pharmacokinetic (PK), metabolism, and routes of excretion of aticaprant and its metabolites in excreta and in plasma after a single oral dose 14C-aticaprant in healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history (screening only), vital signs, and electrocardiogram (ECG) performed at screening and admission to the study site on Day -1. Minor abnormalities in ECG, which are not considered to be of clinical significance by the investigator, are acceptable
* Body weight not less than 50 kilograms (kg) and body mass index (BMI; weight [kg]/height^2 [m^2]) within the range of 18.0 to 29.9 kilogram per meter square (kg/m^2) (inclusive)
* Blood pressure (after the participant is supine for 5 minutes) between 90 millimeters of mercury (mmHg) and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic at screening and Day -1
* A 12-lead ECG consistent with normal cardiac conduction and function, at screening and Day -1, including: sinus rhythm; pulse rate between 40 and 100 beat per minutes (bpm), extremes included; QTc interval less than or equal to (<=) 450 milliseconds (ms) for men; QRS interval of less than (<) 120 ms; PR interval < 210 ms; morphology consistent with healthy cardiac conduction and function
* Non-smokers (not smoked for 3 months prior to screening)

Exclusion Criteria:

* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin, or malignancy, which is considered cured with minimal risk of recurrence)
* Known allergies, hypersensitivity, or intolerance to aticaprant or its excipients
* History of clinically significant (example: in the opinion of the investigator) drug and/or food allergies
* Participant has presence of left bundle branch block, atrioventricular block (second degree or higher), or a permanent pacemaker or implantable cardioverter defibrillator
* Anatomical (nasal) abnormalities which may make the placement of the nasoduodenal tube difficult (only for participants with duodenal sampling)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Plasma Concentrations of Aticaprant and its Metabolite M3 | Up to Day 39
  Plasma samples will be analyzed to determine concentrations of aticaprant and its Metabolite M3 using a validated, specific, and sensitive liquid chromatography (LC)-mass spectrometry (MS)/MS method.
Duodenal Concentrations of Aticaprant and its Metabolite M3 | Pre-dose, 3.75 hour, 4 hour and 5 hour of Day 1
  Duodenal fluid samples will be analyzed to determine concentrations of aticaprant and its Metabolite M3 using a, specific, and sensitive (LC-MS/MS) method.
Urine Concentration of Aticaprant and its Metabolites M3 | Pre-dose up to Day 32
  Urine samples will be analyzed to determine concentrations of aticaprant and its metabolite M3 using a, specific, and sensitive (LC-MS/MS) method.
Total Radioactivity Concentration of 14C-aticaprant in Whole Blood | Pre-dose up to Day 14
  Total radioactivity concentration of 14C-aticaprant in whole blood will be performed via liquid scintillation counting.
Total Radioactivity Concentration of 14C-aticaprant in Plasma | Pre-dose up to Day 14
  Total radioactivity concentration of 14C-aticaprant in plasma will be performed via liquid scintillation counting.
Total Radioactivity Concentration of 14C-aticaprant in Duodenal Fluid | Pre-dose, 3.75 hour, 4 hour and 5 hour of Day 1
  Total radioactivity concentration of 14C-aticaprant in duodenal fluid samples will be performed via liquid scintillation counting.
Amount of Total Radioactivity of 14C-aticaprant in Urine | Up to Day 32
  Amount of total radioactivity of 14C-aticaprant in urine will be performed via liquid scintillation counting.
Amount of Total Radioactivity of 14C-aticaprant in Feces | Up to Day 32
  Amount of total radioactivity of 14C-aticaprant in feces will be performed via liquid scintillation counting.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to Day 67
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Number of Participants with Clinical Laboratory Abnormalities | Up to Day 67
  Number of participants with clinical laboratory abnormalities (including serum chemistry, hematology and urinalysis) will be reported.
Number of Participants with Electrocardiogram (ECG) Abnormalities | Up to Day 67
  Number of participants with ECG abnormalities will be reported.
Number of Participants with Vital Signs Abnormalities | Up to Day 67
  Number of participants with vital signs abnormalities (including body temperature, pulse rate, respiratory rate, blood pressure [systolic and diastolic]) will be reported.
Number of Participants with Physical Examination Abnormalities | Up to Day 67
  Number of participants with physical examination abnormalities will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency